CLINICAL TRIAL: NCT01867086
Title: Phase II Trial of Adjuvant Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Vaccine (FANG™) Integrated With Chemotherapy for Patients With Recurrent Cisplatinum Sensitive Ovarian Cancer Participating in Study CL-PTL 105
Brief Title: Salvage Ovarian FANG™ Vaccine + Carboplatinum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL 110
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer
Keywords: ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vigil™ Vaccine (Experimental): Patients meeting eligibility criteria will receive either carboplatinum alone (AUC 6/30 minute infusion) or carboplatinum (AUC 5/30 minute infusion) and taxol (175 mg/m2 3-hour infusion) one day prior to Vigil™ 1.0 x 10e7 cells/ intradermal injection, once every three weeks. At recurrence, patients allergic to carboplatinum will receive docetaxel 75 mg/m2/1 hour infusion, one day prior to Vigil™ 1.0 x 10e7 cells/intradermal injection every 3 weeks. Patients with stable disease (SD) or better and unable to tolerate continued chemotherapy will be allowed to continue Vigil™ alone for up to 12 cycles or as long as vaccine is available; conversely, patients with SD or better who exhaust Vigil™ supply may continue on chemotherapy alone.
  Interventions: Biological: Vigil™ Vaccine; Drug: Carboplatinum; Drug: Carboplatinum and Taxol

INTERVENTIONS:
Biological: Vigil™ Vaccine — Patients meeting eligibility criteria will receive Vigil™ 1.0 x 10e7 cells/intradermal injection once every 3 weeks.
  Other Names: bi-shRNA furin and GMCSF Augmented Autologous Tumor Cell Vaccine; formerly known as FANG™
Drug: Carboplatinum — Patients meeting eligibility criteria will receive either carboplatinum alone (AUC 6/30 minute infusion) or carboplatinum (AUC 5/30 minute infusion) and taxol (175 mg/m2 3-hour infusion) one day prior to Vigil™ 1.0 x 10e7 cells/ intradermal injection, once every three weeks. At recurrence, patients allergic to carboplatinum will receive docetaxel 75 mg/m2/1 hour infusion, one day prior to Vigil™ 1.0 x 10e7 cells/intradermal injection every 3 weeks. Patients with stable disease (SD) or better and unable to tolerate continued chemotherapy will be allowed to continue Vigil™ alone for up to 12 cycles or as long as vaccine is available; conversely, patients with SD or better who exhaust Vigil™ supply may continue on chemotherapy alone.
Drug: Carboplatinum and Taxol — Patients meeting eligibility criteria will receive either carboplatinum alone (AUC 6/30 minute infusion) or carboplatinum (AUC 5/30 minute infusion) and taxol (175 mg/m2 3-hour infusion one day prior to Vigil™ 1.0 x 10e7 cells/ intradermal injection, once every three weeks. At recurrence, patients allergic to carboplatinum will receive docetaxel 75 mg/m2/1 hour infusion, one day prior to Vigil™ 1.0 x 10e7 cells/intradermal injection every 3 weeks. Patients with stable disease (SD) or better and unable to tolerate continued chemotherapy will be allowed to continue Vigil™ alone for up to 12 cycles or as long as vaccine is available; conversely, patients with SD or better who exhaust Vigil™ supply may continue on chemotherapy alone.

SUMMARY:
This is a Phase II study of Vigil™ autologous tumor cell vaccine integrated with carboplatinum. All patients will have Vigil™ prepared and stored from ovarian tumor cells obtained at the time of primary surgical debulking. Patients meeting eligibility criteria will receive either carboplatinum alone (AUC 6/30 minute infusion) or carboplatinum (AUC 5/30 minute infusion) and taxol (175 mg/m2/3 hour infusion) one day prior to Vigil™ 1.0 x 10e7 cells/intradermal injection, once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed papillary serous or endometrioid ovarian cancer.
2. Previous randomization to Gradalis, Inc. protocol CL-PTL 105; observation arm (Group B) or or patients with vaccine prepared for CL-PTL 105 but did not otherwise qualify.
3. Recurrent cisplatinum-sensitive disease (defined as the appearance of any measurable or evaluable lesion or as asymptomatic CA-125 levels greater than 100 u/mL at two consecutive measurements after a 6 month period after platinum treatment.
4. Successful manufacturing of 4 vials of Vigil™ vaccine.
5. Recovered from all clinically relevant toxicities related to prior therapies.
6. ECOG PS 0-2 prior to Vigil™ vaccine administration.
7. Normal organ and marrow function as defined below:

   1. Absolute granulocyte count ≥ 1,500/mm3
   2. Absolute lymphocyte count ≥ 200/mm3
   3. Platelets ≥ 100,000/mm3
   4. Total bilirubin ≤ 1.5 x ULN
   5. AST(SGOT)/ALT(SGPT)/alkaline phosphatase ≤ 2.5 x ULN
   6. Creatinine < 1.5 mg/dL
8. Patients must be off all "statin" drugs for ≥ 2 weeks prior to initiation of therapy.
9. Ability to understand and the willingness to sign a written informed protocol specific consent.

Exclusion Criteria:

1. Surgery involving general anesthesia, chemotherapy, radiotherapy, steroid therapy, or immunotherapy within 4 weeks prior to vaccination. Chemotherapy within 3 weeks prior to vaccination. Steroid therapy within 1 week prior to vaccination.
2. Patient must not have received any other investigational agents within 4 weeks prior to study entry.
3. Patients who require parenteral hydration of nutrition and have evidence of partial bowel obstruction or perforation.
4. Patients with history of brain metastases.
5. Patients with compromised pulmonary disease.
6. Short term (<30 days) concurrent systemic steroids ≤ 0.25 mg/kg prednisone per day (maximum 7.5 mg/day) and bronchodilators (inhaled steroids) are permitted; other steroid regimens and/or immunosuppressives are excluded.
7. Prior splenectomy.
8. Prior malignancy (excluding nonmelanoma carcinomas of the skin and carcinoma in situ cervix) unless in remission for ≥ 2 years.
9. Kaposi's Sarcoma.
10. Patients with peripheral neuropathy ≥2 (paclitaxel).
11. Uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
12. Patients with known HIV.
13. Patients with chronic Hepatitis B and C infection.
14. Patients with uncontrolled autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minal Barve, MD, Principal Investigator — Principal Investigator
Locations (1):
- Mary Crowley Cancer Research Centers, Dallas, Texas, United States

REFERENCES:
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited subjects from CL-PTL-105 who recurred and were either randomized to the control/observation arm (Group B) or screen-failed but had successful manufacturing of Vigil (minimum of 4 doses).
Pre-assignment Details: 1 subject was enrolled and administered Vigil plus Carboplatinum. This subject did not complete treatment due to disease progression.
Groups:
- Vigil™ Vaccine: Patients meeting eligibility criteria will receive either carboplatinum alone (AUC 6/30 minute infusion) or carboplatinum (AUC 5/30 minute infusion) and taxol (175 mg/m2 3-hour infusion) one day prior to Vigil™ 1.0 x 10e7 cells/ intradermal injection, once every three weeks. At recurrence, patients allergic to carboplatinum will receive docetaxel 75 mg/m2/1 hour infusion, one day prior to Vigil™ 1.0 x 10e7 cells/intradermal injection every 3 weeks. Patients with stable disease (SD) or better and unable to tolerate continued chemotherapy will be allowed to continue Vigil™ alone for up to 12 cycles or as long as vaccine is available; conversely, patients with SD or better who exhaust Vigil™ supply may continue on chemotherapy alone.
  Vigil™ Vaccine: Patients meeting eligibility criteria will receive Vigil™ 1.0 x 10e7 cells/intradermal injection once every 3 weeks.
  Carboplatinum: Patients meeting eligibility criteria will receive either carboplatinum alone (AUC 6/30 minute infusion)
Period: Overall Study
Arm/Group | Vigil™ Vaccine
Started | 1
Completed | 0 ("Completed" means subject had been given all manufactured doses.)
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Vigil™ Vaccine: Patients meeting eligibility criteria will receive either carboplatinum alone (AUC 6/30 minute infusion) or carboplatinum (AUC 5/30 minute infusion) and taxol (175 mg/m2 3-hour infusion) one day prior to Vigil™ 1.0 x 10e7 cells/ intradermal injection, once every three weeks.
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) will be determined following Carboplatinum integrated with Vigil vaccine in patients failing standard of care in study CL-PTL 105 or in those not otherwise qualifying after vaccine production. This will be measured from the treatment start date (date of first dose) to either the date the patient is first recorded as having disease recurrence (even if the patient went off treatment because of toxicity), or the date of death if the patient dies due to any causes before progression.
Time Frame: 24 months
Population: 1 subject was enrolled and started Vigil treatment plus Carboplatinum. This subject did not complete treatment due to disease progression. There is no Outcome Measure Data table because Time to Progression (TTP) and Response Rate (RR) were not collected and analyzed. This study was terminated.
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 0

2. Primary Outcome: Response Rate
Description: Response will be evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline.
Time Frame: Up to 12 months
Population: as for outcome 1
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 0

3. Secondary Outcome: Immune Analysis in Blood
Description: To determine if subjects will have a positive (defined as >10 ELISPOTS from baseline) immune response to Vigil. Blood was collected to compare ELISPOT results from baseline until 30 days after last dose.
Time Frame: Baseline, End of Treatment (30 days after last dose) up to 12 months
Population: 1 subject was enrolled and started Vigil treatment plus Carboplatinum. This subject did not complete treatment due to disease progression. After 12 months, subject had positive ELISPOT response. Statistical analysis was not done. This study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 1
Participants
  ELISPOT-Positive After 12 months | 1
  ELISPOT-Negative After 12 months | 0

4. Other Pre Specified Outcome: Number of Alive Subjects
Description: Survival status of patients after treatment will be determined.
Time Frame: 24 months
Population: 1 subject was enrolled and started Vigil treatment plus Carboplatinum. This subject did not complete treatment due to disease progression. After 24 months, subject was not alive. Statistical analysis was not done. This study was terminated.
Measure: Count of Participants; unit: Participants
Arm/Group | Vigil™ Vaccine
Number analyzed (Participants) | 1
Participants
  Alive Subjects After 24 months | 0
  Dead Subjects After 24 months | 1

ADVERSE EVENTS:
Arm/Group | Vigil™ Vaccine
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vigil™ Vaccine (N=1)
Injection Site Reaction (General disorders) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes